CLINICAL TRIAL: NCT03581617
Title: Prognostic Markers in Women With Primary Unexplained Infertility
Brief Title: Infections and Unexplained Infertility
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Giuseppe Lo Monte, Doctor, University Hospital of Ferrara
Other Study IDs: PRUAlGR-2013-00000084
Record Dates: First submitted 2018-06-04; First posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Infertility, Female
Keywords: Infertility; NK cells; HLA-G
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infertile women: Inclusion criteria for the study group will be as follows: 21-38 years old, primary infertility (no live birth), regular menstrual cycle (24-35 days), body mass index (BMI) ≤ 25, FSH <10 mUI/mL, E2 < 50 pg/ml on day 2-3 of the menstrual cycle. They will be recruited at admission for tubal patency assessment.
  Interventions: Diagnostic Test: NK cell analysis; Diagnostic Test: Herpesvirus detection; Diagnostic Test: sHLA-G analysis; Diagnostic Test: HLA-G 14bp INS/DEL typing; Diagnostic Test: sHLA-E analysis
- Fertile women: Inclusion criteria for control group will be as follows: 21-35 years old, almost one live birth, regular menstrual cycle (24-35 days), BMI ≤ 25, FSH <10 mUI/mL, E2 < 50 pg/mL on day 2-3 of the menstrual cycle. Women with endometritis, endometriosis, tubal factor, ovulatory dysfunction, anatomical uterine pathologies will be excluded.
  Interventions: Diagnostic Test: NK cell analysis; Diagnostic Test: Herpesvirus detection; Diagnostic Test: sHLA-G analysis; Diagnostic Test: HLA-G 14bp INS/DEL typing; Diagnostic Test: sHLA-E analysis

INTERVENTIONS:
Diagnostic Test: NK cell analysis — We selected to perform the study during the proliferative phase (day 9-11), where only resident eNK cells are present in the endometrium. The samples will be analyzed with the following methods, that are routinely used in the OUs of the proposal:
  - pNK cell analysis: PBMCs will be purified with Ficoll solution and NK cells will be analyzed by flow cytometry (FacsVantage, BD) with anti-CD56, CD16, CD9, CD49a, KIRs, LILRB1, LILRB2, CD94, CD107a eNK cell analysis: eNK cells will be obtained from endometrial biopsies during proliferative phase, determined by ultrasound scan and analyzed for NK cell subtypes and KIRs, LILRB1, LILRB2, CD94, CD107a expression by flow cytometry
Diagnostic Test: Herpesvirus detection — Herpesvirus detection: DNA will be analyzed by specific primers for HSV-1, HSV-2, EBV, CMV, HHV-6, HHV-7, VZV, and HHV-8, with PCR and nested PCR
Diagnostic Test: sHLA-G analysis — sHLA-G analysis: sHLA-G quantification in plasma and endometrial flushing will be performed by ELISA using anti-HLA-G (G233) and anti-beta2-microglobulin HRP-conjugated moAbs (Exbio)
Diagnostic Test: HLA-G 14bp INS/DEL typing — Genomic DNA will be genotyped by RealTime PCR
Diagnostic Test: sHLA-E analysis — sHLA-E analysis: sHLA-E quantification in plasma and endometrial flushing will be performed by ELISA using anti-HLA-E (3D12, eBioscience) and anti-beta2-microglobulin HRP-conjugated moAbs (Exbio)

SUMMARY:
1. Background: In women, unexplained infertility has been associated with a range of cellular and molecular defects in the endometrium, adverse immune responses and immunological factors. Natural killer (NK) cells are included as they constitute the most abundant leukocyte population in the decidua. While decidua NK cells were extensively investigated, the study of endometrial eNK cells still lacks comprehensive researches. The reduction in eNK frequency has been associated with infertility status, in particular in the presence of a concomitant herpesvirus viremia. Since herpesviruses use as immune-escape HLA-G and HLA-E molecules, that are immune-inhibitory and important for a correct placentation, they could represent infertility co-factors.
2. Aims: Since lack of an accurate diagnosis in reproductive medicine leads to treatment failure, this proposal focuses on eNK cell characterization as a diagnostic factor for unexplained women infertility. We will evaluate also co-factors, taking into consideration herpesvirus infection and HLA-G and HLA-E expression.
3. Methods: Peripheral blood and endometrial NK cells will be immune-phenotyped and cell count and activation status (CD107a, IL-6, IL-10, IL-17) will be correlated with infertility condition. The implication of herpesvirus will be evaluated by DNA from peripheral blood and endometrial flushing samples analysis by HSV-1, HSV-2, EBV, CMV, HHV-6, HHV-7, VZV and HHV-8 specific primers an PCR technique. HLA-G and HLA-E expression will be analyzed in peripheral blood and endometrial environment by flow cytometry and ELISA tests and correlated by NK cell expression of their receptors (KIRs, LILRB1/2, NKG2A).
4. Expected results: On the basis of our preliminary results, we expect to identify NK cells as prognostic marker for primary unexplained infertility, with herpesvirus infection and HLA-G and HLA-E expression as co-factors. These data will be of importance in the management of infertile women.

DETAILED DESCRIPTION:
Primary Objective The main challenge of this project is to define the potential role of NK cells as a prognostic marker for primary unexplained infertility. To achieve this objective we will perform a prospective study on a cohort of 100 unexplained infertile women. Peripheral blood and endometrial NK cells will be immune phenotyped and their activation status will be analyzed. Meanwhile, the presence of herpesvirus infection will be evaluated in peripheral blood and correlated with the results of NK analysis. These data will clarify the role of NK cells in infertile female conditions, evaluating the implication of herpesvirus infection as a cofactor for NK cell status. These data will provide a proof of principle of the use of NK cell analysis as a predictive marker for unexplained infertility.

Secondary Objective The secondary objective is to evaluate the mechanisms at the basis of the NK cell status in infertility. Since HLA-G and HLA-E expression is modified by herpesvirus infection (9), as an immune escape mechanism, and these antigens are responsible of a correct embryo implantation (14), we will analyze the levels of these molecules in peripheral blood and endometrial environment. Meanwhile, HLA-G and HLA-E genetic polymorphisms will be analyzed. These results will be correlated with the presence of herpesvirus infection, KIR, LILRB and NKG2A receptor expression on pNK and eNK cells. These data will clarify the implication of HLA-G and HLA-E expression and genetic background in the control of NK cell activation and herpesvirus infection in infertile women.

The achievement of these objectives will be obtained with 6 workpackages/aims (WP)

1. Infertile women characterization (WP1) (1-20mth) We will recruit 100 unexplained infertile women and 30 control women. These women will be clinically evaluated, establishing a clinical database. From each woman, we will obtain peripheral blood samples, endometrium biopsies, and uterine flushing.
2. NK cell immune-phenotype (WP2) (1-20mth) NK cells from peripheral blood and endometrium will be analyzed for subtype percentages (CD56, CD16, CD9, CD49a), and for the expression of KIR, LILRB-1 and -2 and CD94/NKG2A receptors, that are known to interact with HLA-G and HLA-E molecules producing inhibitory signals.
3. Th1, Th2, Th17 and LIF (WP3). (1-20 mth) Th1, Th2, Th17 and LIF levels will be analyzed in plasma and uterine flushing samples, to evaluate activation status. The results will be correlated with NK cell count.
4. Herpesvirus infection (WP4) (12-24mth) Herpesvirus DNA (HSV-1, HSV-2, EBV, CMV, HHV-6, HHV-7, VZV and HHV-8) presence will be analyzed in peripheral blood and uterine flushing.
5. HLA-G (WP5) (12-24mth) HLA-G molecules are expressed as both membrane (HLA-G1) and soluble (HLA-G5, from mRNA alternative splicing; sHLA-G1, from membrane shedding) molecules. The expression of the membrane and soluble HLA-G will be evaluated in peripheral blood and endometrium. HLA-G expression is controlled by a polymorphism of insertion/deletion (ins/del) of 14 base pairs (rs66554220), where the deletion of 14bp stabilizes the mRNA producing higher levels of HLA-G (15). We will genotype the women for rs66554220 polymorphism, to evaluate the implication in HLA-G levels of expression in infertile condition.
6. HLA-E (WP6) (12-24mth) HLA-E molecules are expressed as both membrane and soluble molecules. The expression of the membrane and soluble HLA-E will be evaluated in peripheral blood and endometrium. Two non-synonymous alleles of HLA-E have been identified, HLA-ER (E*0101) and HLA-EG (E*0103) (16), where HLA-E expression of the EG protein was higher than ER. We will genotype the women for HLA-E polymorphisms, to evaluate the implication in infertility.

ELIGIBILITY:
Inclusion criteria for the study group :

* 21-38 years old,
* primary infertility (no live birth),
* regular menstrual cycle (24-35 days),
* body mass index (BMI) ≤ 25, FSH <10 mUI/mL,
* E2 < 50 pg/ml on day 2-3 of the menstrual cycle. Recruitment at admission for tubal patency assessment.

Inclusion criteria for control group:

* 21-35 years old,
* almost one live birth,
* regular menstrual cycle (24-35 days),
* BMI ≤ 25, FSH <10 mUI/mL,
* E2 < 50 pg/mL on day 2-3 of the menstrual cycle

Exclusion criteria:

* endometritis,
* endometriosis,
* tubal factor,
* ovulatory dysfunction,
* anatomical uterine pathologies.

Ages: 21 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Infertile women
Study Population: This will be a prospective non-interventional clinical study, based on biological specimens sampled during current standard clinical practice. Based on our preliminary results, we will enroll 100 infertile and 30 control women to achieve a 0.8 power with 5% alpha error in detecting differences between infertile and fertile women.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2015-11-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Prognostic value of NK cells in female idiopathic infertility | 20 months
  Percentage of (e)NK CD56brightCD16-
Herpesvirus detection | 16 months
  Presence of HHVs infection in endometrial cells

SECONDARY OUTCOMES:
Levels of sHLA-G and sHLA-E cellule pNK e eNK | 16 months
  Levels of sHLA-G and sHLA-E in uterine flushing samples
HLA-G and HLA-E genetic polymorphisms | 10 months
  Frequency of HLA-G and HLA-E genetic polymorphisms
Cytokines levels in endometrial flushing samples | 10 months
  Levels of Th1 and Th2 cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Lo Monte, M.D., Principal Investigator — Università di Ferarra

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rizzo R, Lo Monte G, Bortolotti D, Graziano A, Gentili V, Di Luca D, Marci R. Impact of soluble HLA-G levels and endometrial NK cells in uterine flushing samples from primary and secondary unexplained infertile women. Int J Mol Sci. 2015 Mar 10;16(3):5510-6. doi: 10.3390/ijms16035510. PMID 25764161